CLINICAL TRIAL: NCT00841984
Title: Evaluation of in Vitro NMR Spectroscopy to Identify Inborn Errors of Metabolism in Patients With Complex Neurological Diseases
Brief Title: In Vitro NMR Spectroscopy in Neurological Diseases
Acronym: SPECMET
Status: Terminated | Type: Observational
Why Stopped: not enough enrollment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Zakia Idir, Department Clinical Research
Other Study IDs: P051057
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Neurological Diseases
Keywords: Magnetic resonance spectroscopy; neurological diseases; metabolic; inborn errors of metabolism; Complex neurological diseases of unknown cause
MeSH Terms: conditions — Metabolism, Inborn Errors

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urines, cerebrospinal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: patients with complex neurological disease of unknown cause
- 2: positive controls : patients with already known metabolic disease for whom we already have CSF or urines
- 3: negative controls: patients with non metabolic neurological disorders of known cause hospitalized for a lumbar puncture

SUMMARY:
The search for metabolic abnormalities in patients with neurological disorders represents an important challenge 1) to identify new potentially treatable inherited metabolic diseases, and 2) to identify biomarkers or new treatments in more common neurodegenerative or neurogenetic disorders.

This approach is currently limited by the fact that techniques aiming at identifying abnormal metabolites in human fluids (metabolomics) only detect subsets of molecules and that no general assays is available to detect abnormalities in the metabolism of complex molecules that takes place within cell organelles. As a consequence, only limited parts of the metabolism can be studied simultaneously.

The aim of this study is to evaluate whether NRM spectroscopy of body fluids (urines, cerebrospinal fluid) could allow to detect new metabolic abnormalities in patients with complex neurological diseases.

DETAILED DESCRIPTION:
It is now established that most inborn errors of metabolism may present in adulthood as a neurological disorder. The diagnosis of these diseases is essential because, unlike the so-called neurodegenerative diseases, metabolic diseases are often accessible to specific treatments.

Conversely, many patients are followed for a complex neurological disease of unknown cause. We hypothesize that a significant proportion of these patients carry yet undetected inborn error of metabolism.

Recently, the use of Nuclear magnetic resonance spectroscopy (NMRS) has uncovered new metabolic diseases leading sometimes to specific treatments. However, the place of this technique in the investigation of patients with complex neurological diseases remains to be determined.

The primary goal of this project is to assess the interest of NMRS in urine and CSF to search metabolic abnormalities, not detected by conventional biochemical techniques. It is an open study. The study will be conducted in close collaboration between the neurology and genetic departments of the Pitié-Salpêtrière hospital, on the one hand and the nuclear medicine department of Poitiers in the other. 250 patients will be included over a period of 2-3 years and will be divided into 4 groups: Group 1: patients with complex neurological disease of unknown cause (200 patients) for whom urines and CSF will be collected. Group 2: positive controls (25 patients): patients with already known metabolic disease for whom we already have CSF or urines. Group 3: negative controls (25 patients): patients with non metabolic neurological disorders of known cause hospitalized for a lumbar puncture.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Any patient with an unexplained complex neurological disease
* Group 2: Patients with known inborn error of metabolism
* Group 3: patients with known non metabolic disease

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with an unexplained complex neurological disease
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2006-07; Primary Completion 2008-07 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with new metabolic diseases | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Sedel, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Neurology department, Pitié-Salpêtrière Hospital, Paris, France